CLINICAL TRIAL: NCT03753854
Title: Effects of Obstructive Sleep Apnea on the Frequency of Vaso-occlusive Crises Events and Bio-physical Markers in Sickle Cell Disease
Brief Title: Sleep Apnea in Sickle Cell Disease
Acronym: DREPAPNEE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL17_0784; 2017-A03352-51 (Other: ANSM number)
Record Dates: First submitted 2018-11-20; First posted 2018-11-27 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; obstructive sleep apnoea; vaso-occlusive crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Sleep Apnea, Obstructive; Vaso-Occlusive Crises | interventions — Polysomnography; Blood Specimen Collection; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SS patients (Active Comparator): Homozygous sickle cell patients
  Each patient will undergo the following:
  1. polysomnography and oxygen saturation exam
  2. calculation of VOC rate within the two previous years
  3. Blood samples
  4. Physiological measurements
  Interventions: Diagnostic Test: polysomnography and oxygen saturation exam; Biological: calculation of VOC frequency between the first polysomnography and the end of the first year of continuous positive airway pressure treatment; Biological: Blood samples; Other: Physiological measurements
- SS patients apneic (Experimental): Homozygous sickle cell patients after one year of continuous positive airway pressure treatment
  Each patient will undergo the following:
  1. polysomnography and oxygen saturation exam
  2. calculation of VOC rate within the two previous years
  3. Blood samples
  4. Physiological measurements
  Interventions: Diagnostic Test: polysomnography and oxygen saturation exam; Biological: calculation of VOC frequency between the first polysomnography and the end of the first year of continuous positive airway pressure treatment; Biological: Blood samples; Other: Physiological measurements; Other: Continuous Positive Airway Pressure

INTERVENTIONS:
Diagnostic Test: polysomnography and oxygen saturation exam — Measurement of the Apnea/hypopnea index (AHI) and oxygen saturation
Biological: calculation of VOC frequency between the first polysomnography and the end of the first year of continuous positive airway pressure treatment — calculation of VOC rate within the two previous years or between first polysomnography and one year of continuous positive airway pressure treatment
Biological: Blood samples — Blood samples with measurements of hematological, hemorheological, inflammatory and blood coagulation markers
Other: Physiological measurements — Evaluation of microvascular reactivity and autonomic nervous system activity
Other: Continuous Positive Airway Pressure — Continuous Positive Airway Pressure during 1 year
  Arms: SS patients apneic

SUMMARY:
Despite the fact that obstructive sleep apnoea (OSA) is highly prevalent in the sickle cell population, studies focusing on the associations of the two diseases and their common pathophysiological mechanisms are scarce. OSA is one of the most common conditions responsible for hemoglobin desaturation. The nocturnal hemoglobin desaturation occurring in some sickle cell disease (SCD) patients with OSA could trigger hemoglobin S polymerization and red blood cell (RBC) sickling, leading to further blood rheological alterations, hence increasing the risks for VOC. Moreover, OSA has been demonstrated to increase oxidative stress and inflammation in non Sickle Cell Disease (SCD) patients, which, in SCD patients, could increase the risk for complications. Finally, OSA is accompanied by impaired vascular function and autonomic nervous system dysfunction in the general population. Indeed, the presence of OSA in SCD could increase the clinical severity of patients and the frequency of VOC.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous HbS (Hemoglobin S) (SS) patients,
* aged between 15 and 3 months and 50 years old,
* in steady state (i.e. without vaso-occlusive crisis or recent blood transfusion),
* followed by the sickle cell center of the Hospices Civils de Lyon,
* and showing symptoms of OSA.

Exclusion Criteria:

* Patients receiving treatment of OSA,
* recent blood transfusion (less than 2 months),
* patients not at steady state (VOC or acute chest syndrome less than 2 months),
* pregnancy.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
number of VOC crises required hospitalization in the previous two years | day 1
  Calculated over a 2 years period before inclusion. VOC requiring hospitalizations will be recorded.
  Measured at day 1

SECONDARY OUTCOMES:
Blood inflammatory markers | An average of 1 month
  Blood inflammatory markers : C Reactive Protein (CRP, mg/L) The morning after the polysomnography blood samples will be collected (M1 +/- 15 days)
Blood inflammatory markers | Day 365
  Blood inflammatory markers : C Reactive Protein (CRP, mg/L)
Markers of blood coagulation | An average of 1 month
  Biological risk factors of VOC : prothrombin time (PT, s), D-dimer (µg/L), Fibrinogen (g/L), Activated Thromboplastin Time (APPT, s), protein C and protein S (%) The morning after the polysomnography blood samples will be collected (M1 +/- 15 days)
Markers of blood coagulation | Day 365
  prothrombin time (PT, s), D-dimer (µg/L), Fibrinogen (g/L), Activated Thromboplastin Time (APPT, s), protein C and protein S (%)
Blood cell counts and markers of hemolysis | An average of 1 month
  Biological risk factors of VOC : Blood cell counts and markers of hemolysis : red blood cell count (G/L), neutrophil count (G/L), hemoglobin concentration (g/dL), hematocrit (%), mean corpuscular volume (MCV, fl), mean corpuscular hemoglobin concentration (MCHC, pg), platelet count (G/L), lactate dehydrogenase (LDH, IU), bilirubin (µg/L), aspartate transaminase (AST, U/L).
  The morning after the polysomnography blood samples will be collected (M1 +/- 15 days)
Blood cell counts and markers of hemolysis | Day 365
  Blood cell counts and markers of hemolysis : red blood cell count (G/L), neutrophil count (G/L), hemoglobin concentration (g/dL), hematocrit (%), mean corpuscular volume (MCV, fl), mean corpuscular hemoglobin concentration (MCHC, pg), platelet count (G/L), lactate dehydrogenase (LDH, IU), bilirubin (µg/L), aspartate transaminase (AST, U/L).
Markers of nitric oxide metabolism | An average of 1 month
  Biological risk factors of VOC : markers of nitric oxide production nitrites, nitrate, nitrotyrosine The morning after the polysomnography blood samples will be collected (M1 +/- 15 days)
Markers of nitric oxide metabolism | Day 365
  markers of nitric oxide production nitrites, nitrate, nitrotyrosine
Oxidative stress markers | An average of 1 month
  Biological risk factors of VOC : protein oxidation marker (advanced oxidation protein products), markers of lipid peroxidation (malondialdehyde), antioxidant enzymatic activities (super oxide dismutase, catalase, glutathione peroxidase), antioxidant power (ferric reducing ability of plasma) The morning after the polysomnography blood samples will be collected (M1 +/- 15 days)
Oxidative stress markers | Day 365
  protein oxidation marker (advanced oxidation protein products), markers of lipid peroxidation (malondialdehyde), antioxidant enzymatic activities (super oxide dismutase, catalase, glutathione peroxidase), antioxidant power (ferric reducing ability of plasma)
Hemorheological parameters | An average of 1 month
  blood viscosity (cP) measured with a cone plate viscometer at several shear rates, red blood cell deformability (a.u) measured by ektacytometry at several shear stresses, red blood cell aggregation (%) properties measured by laser backscatter method.
  The morning after the polysomnography blood samples will be collected (M1 +/- 15 days)
Hemorheological parameters | Day 365
  Biological risk factors of VOC : blood viscosity (cP) measured with a cone plate viscometer at several shear rates, red blood cell deformability (a.u) measured by ektacytometry at several shear stresses, red blood cell aggregation (%) properties measured by laser backscatter method.
Arterial blood gases | An average of 1 month
  Biological risk factors of VOC : oxygen and carbon dioxide pressure (mmHg), pH The morning after the polysomnography blood samples will be collected (M1 +/- 15 days)
Arterial blood gases | Day 365
  oxygen and carbon dioxide pressure (mmHg), pH
Vascular function (microvascular reactivity to skin heating test) | Day 1
  Physiological risk factors of VOC : A laser Doppler flowmeter (Periflux 5000 Perimed) will be used to measure skin blood flow in resting condition and during a local thermal hyperemia (LTH) test (temperature will be increased from 33 °C to 42 °C) for 35 min. The peak response during the LTH reflects vasodilatation caused by axonal reflex while the delayed plateau response of the LTH test is mainly dependent on the ability to produce nitric oxide to promote vasodilation.
Vascular function (microvascular reactivity to skin heating test) | Day 365
  A laser Doppler flowmeter (Periflux 5000 Perimed) will be used to measure skin blood flow in resting condition and during a local thermal hyperemia (LTH) test (temperature will be increased from 33 °C to 42 °C) for 35 min. The peak response during the LTH reflects vasodilatation caused by axonal reflex while the delayed plateau response of the LTH test is mainly dependent on the ability to produce nitric oxide to promote vasodilation.
autonomic nervous system activity (measured by heart rate variability analysis) | Day 1
  Physiological risk factors of VOC : electrocardiographic signals acquired by the polysomnographic machine will be extracted and the R-R intervals will be used for time domain spectral analyses to calculate several indices reflecting the activity of the autonomic nervous system activity. The ratio between the low frequency and the high frequency powers (LF/HF) will be used to characterize the autonomic imbalance.
autonomic nervous system activity (measured by heart rate variability analysis) | Day 365
  electrocardiographic signals acquired by the polysomnographic machine will be extracted and the R-R intervals will be used for time domain spectral analyses to calculate several indices reflecting the activity of the autonomic nervous system activity. The ratio between the low frequency and the high frequency powers (LF/HF) will be used to characterize the autonomic imbalance.
Frequency of VOC | Day 365
  Number of VOC requiring hospitalizations during the past year

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Edouard Herriot, Lyon
  - Centre Léon Berard, Lyon
  - Hôpital de la Croix Rousse, Lyon

REFERENCES:
- [Derived] Stauffer E, Poutrel S, Cannas G, Gauthier A, Fort R, Bertrand Y, Renoux C, Joly P, Boisson C, Hot A, Peter-Derex L, Pialoux V, PetitJean T, Connes P. Nocturnal Hypoxemia Rather Than Obstructive Sleep Apnea Is Associated With Decreased Red Blood Cell Deformability and Enhanced Hemolysis in Patients With Sickle Cell Disease. Front Physiol. 2021 Sep 24;12:743399. doi: 10.3389/fphys.2021.743399. eCollection 2021. PMID 34630163